CLINICAL TRIAL: NCT05132738
Title: Ripretinib Used for Preoperative Treatment of Potentially Resectable Locally Advanced and Recurrent Metastatic GIST After Failure of Imatinib Therapy: An Exploratory Study
Brief Title: Ripretinib Used for Resectable Metastatic GIST After Failure of Imatinib Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Hui Cao, Professor, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ripretinib for GIST
Record Dates: First submitted 2021-09-15; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; Ripretinib; Imatinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ripretinib treatment group (Experimental)
  Interventions: Drug: Ripretinib treatment

INTERVENTIONS:
Drug: Ripretinib treatment — Ripretinib: 4-week (28-day) cycle of oral administration of 150 mg q.d. For patients who completed up to 6 consecutive treatment cycles in a the clinical investigator decided whether to perform the operation or not, the specific time and other matters.
  The above medications can be adjusted according to the adverse reactions of subjects according to the protocol at the investigator's discretion. Subjects will continue treatment until disease progression, intolerable toxicity, withdrawal of informed consent, or discontinuation of treatment as judged by the investigator, and the investigator will decide whether to perform early surgery or subsequent treatment regimen.

SUMMARY:
To explore the efficacy and safety of preoperative treatment of potentially resectable locally advanced or recurrent metastatic gastrointestinal stromal tumor (GIST) after failure of treatment.

DETAILED DESCRIPTION:
This study is a single-arm, single-center, exploratory study. A total of 20 patients were enrolled. The patient was orally administered with 150 mg of ripretinib daily. The study is expected to enroll the first patient in August 2021, last patient before March 30, 2023 and end the trial in November 2023. Subjects will receive up to 6 cycles of treatment before surgery, which will occur 1 week after the last dose of study drug. The subject requires discontinuation of study treatment or withdrawal from the study due to disease progression, intolerable toxicity, or Investigator's judgment.

The study will be divided into 3 periods: screening period, treatment period (visit period) and follow-up period. All subjects in the study were required to meet all inclusion criteria and exclusion criteria.

In this study, the screening period did not exceed 28 days, and eligible subjects who completed the screening tests and assessments entered the treatment period for study treatment and visits as specified in the protocol. Thereafter, participants entered the follow-up period. The safety follow-up period begins with 30 days of study treatment until 90 days after dosing, and subjects should receive telephone assessments every 30 days. After the safety follow-up period, subjects entered the survival follow-up period. Survival follow-up will be performed every 3 months until 1 year after treatment. Survival information and subsequent treatment information can be collected by effective means such as telephone follow-up. For subjects without radiographic evidence of disease progression, radiographic assessments should continue to be performed at the frequency of efficacy evaluations specified for this study.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be enrolled in the study:

1. Patients voluntarily, and signed a written informed consent, good compliance with follow-up;
2. 18 years ≤ age < 75 years, male or female;
3. Histopathological examination confirmed the diagnosis of gastrointestinal stromal tumors, and immunohistochemical detection of CD117 and/or DOG-1 positive;
4. According to the modified RECISTv1.1-GIST-specific (hereinafter referred to as"mRECIST") criteria, the subject has at least one measurable lesion (the long diameter of non-lymph node lesions is ≥ 1.0 cm or ≥ 2 times the scanning slice thickness); the lesions with definite progression after local treatment can also be considered as measurable lesions; the imaging results must be obtained within 21 days before the first dose;
5. Potentially resectable locally advanced or recurrent metastatic gastrointestinal stromal tumors who have failed imatinib treatment:

   * The number of evaluable lesions is ≤ 5 as judged by CT/MRI;
   * The resection is considered to have significant risks by MDT assessment (meeting any of the following):

     1. The maximum diameter of a single lesion is ≥ 10 cm;
     2. Organ function damage surgery is required (gastrectomy, total gastrectomy, hepatectomy residual liver body ≤ 50% of the normal liver volume);
     3. Multiple organ resection surgery is required (partial gastrectomy combined with pancreatectomy/splenectomy, pancreaticoduodenectomy and abdominoperineal resection);
6. The ECOG physical status score of patients is 0-2;
7. Good organ function and bone marrow reserve, including:

   * Neutrophil count ≥ 1.5 × 109/L
   * Hemoglobin ≥ 90 g/L
   * Platelets ≥ 100 × 109/L
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * AST and ALT ≤ 3 × ULN, and ≤ 5 × ULN in the presence of liver metastases
   * Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (calculated according to Cockcroft-Gault formula)
   * Prothrombin time (PT), international normalized ratio (INR) and partial thromboplastin time ≤ 1.5 × ULN.
   * QTc ≤ 450 ms (male), 470 (female): LVEF ≥ 50%
8. Non-surgically sterilized or female patients of childbearing age need to use a medically recognized contraceptive (such as intrauterine device, contraceptives or condoms) during study treatment and within 90 days after the end of study treatment; non-surgically sterilized female patients of childbearing age need to confirm that they are not pregnant; and must be non-lactating; for male patients with partners of childbearing age, effective regimen contraception should be used during study treatment and within 90 days after the end of study treatment.

Exclusion Criteria:

Patients with any of the following will not be enrolled in the study:

1. Patients with other serious complications who cannot tolerate surgery: such as severe cardiopulmonary disease, heart function below clinical class 2, pulmonary infection, moderate to severe COPD, chronic bronchitis, severe diabetes and/or renal insufficiency, severe hepatitis and/or Child-pugh class C or B whose symptoms are significantly difficult to correct, severe malnutrition, etc.;
2. Occurrence of bleeding, perforation, obstruction and other disease-related complications, requiring emergency surgery;
3. Patients with severe mental illness;
4. The patient has participated in or is participating in other clinical studies , or is taking other TKI agents; has any clinically significant concurrent medical condition such as uncontrolled pulmonary disease, active infection, or any other condition that, in the opinion of the investigator, may affect patient compliance, interfere with interpretation of study results, or expose the patient to safety risks.
5. Active viral infections such as human immunodeficiency virus, hepatitis B, and hepatitis C
6. Pregnant or lactating female patients or patients expecting to become pregnant during study treatment
7. Known hypersensitivity to any component of the study drug.
8. Gastrointestinal abnormalities, including but not limited to:

   * Inability to swallow study drug
   * Malabsorption syndrome
   * Need for intravenous nutrition
9. Any active bleeding, excluding hemorrhoids or gingival bleeding. Has any clinically significant concurrent medical condition, such as uncontrolled pulmonary disease, active infection, or any other condition that, in the opinion of the investigator, may affect patient compliance, interfere with interpretation of study results, or expose the patient to safety risks.
10. The investigator considers that there are other factors that may affect the study results or cause the study to be terminated, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring concomitant treatment, severe laboratory abnormalities, with family or social factors that may affect the safety of patients.
11. Other patients who may affect the conduct of the clinical study in the judgment of the investigator, may be unable to comply with the agreement or unable to cooperate, patients with study risks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
No Evidence of Disease Rate (NED Rate) | baseline
  The primary study endpoint is to investigate the disease-free status rate of ripretinib for the preoperative treatment of potentially resectable locally advanced or recurrent metastatic GIST (NED Rate defined as patients who achieve R0 resection or complete response or macroscopic complete ablation of all known tumor lesions based on imaging assessment, with known tumor lesions assessed by CT or MRI at baseline and within 14 days after surgery, respectively).
No Evidence of Disease Rate (NED Rate) | within 14 days after surgery
  The primary study endpoint is to investigate the disease-free status rate of ripretinib for the preoperative treatment of potentially resectable locally advanced or recurrent metastatic GIST (NED Rate defined as patients who achieve R0 resection or complete response or macroscopic complete ablation of all known tumor lesions based on imaging assessment, with known tumor lesions assessed by CT or MRI at baseline and within 14 days after surgery, respectively).

SECONDARY OUTCOMES:
R0/R1 resection rate | 1 days after surgery
  R0 is the proportion of patients with no microscopic residual after resection/R1 is the proportion of patients with microscopic residual.
Surgery rate | up to 6 months
  The proportion of patients who can undergo surgery.
Objective response rate (ORR) | up to 24 months
  The proportion of patients who achieve complete response and partial response.

OTHER OUTCOMES:
Recurrence-free survival (RFS) | until the date of first documented progression, assessed up to 24 months
  The recurrence-free survival (RFS, defined as the time from initial surgery to the earliest evidence of recurrence) of potentially resectable locally advanced or recurrent metastatic GIST treated with preoperative therapy failure.
Overall survival (OS) | until the date of death from any cause, assessed up to 24 months
  Overall survival (OS, defined as the time from randomization to death from any cause)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Cao, Professor, Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China